CLINICAL TRIAL: NCT07099469
Title: A Randomized Pilot Study of ICNB With Ropivacaine Versus ICNB With Cryotherapy for Postoperative Pain Management After RATS Anatomical Resection for Lung Cancer.
Brief Title: Compairing R-ICNB and C-ICNB for Postoperative Pain Management After Minimal-invasive Anatomical Lung Resection
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Jeroen Hendriks, Prof. Dr. J. Hendriks, University Hospital, Antwerp
Other Study IDs: 004017
Record Dates: First submitted 2025-03-21; First posted 2025-08-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain Management; RATS Surgery
Keywords: C-ICNB; R-ICNB; RATS Surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- R-ICNB: At the end of the procedure, an intercostal block is placed by injecting a local anesthetic into the site of surgery.
- C-ICNB: At the end of the surgery single shot cryotherapy will be placed at 6 levels (T3-T8) with the AtriCure"s cryoICE cryosphere cryoablation probes.

SUMMARY:
This is a pilot study in which a total of 6 people will participate. This study aims to optimize the postoperative pain management of an anatomically minimally invasive lung resection (RATS) by comparing 2 pain-relieving techniques. As standard, an intercostal block is placed at the end of the procedure by injecting a local anesthetic at the site where the patient will be operated on. This study compares the previous method with the use of cryotherapy as an intercostal block. This technique uses cryo probes and blocks postoperative pain for 1-3 months. By comparing both techniques, it is examined whether cryotherapy requires less pain medication and is therefore more effective.

DETAILED DESCRIPTION:
Adequate pain control after robotic-assisted thoracic surgery (RATS) for lung resection is important to improve postoperative mobilisation and recovery, and to prevent postoperative pulmonary complications.

Thoracic epidural analgesia (TEA) is the usual care for postoperative pain management following thoracic surgery. Although the analgesic effect of TEA is clear, failure rates are 9-30% [1, 2, 3] and awake placement is stressful for patients. In addition, TEA is associated with patient immobilisation, bladder dysfunction and hypotension [4]. Based on the best available evidence and the recent guidelines by the Enhanced Recovery After Surgery (ERAS) society, the European Society of Thoracic Surgeons (ESTS) includes early mobilisation after surgery as one of their key recommendations [5]. The department of Thoracic Surgery of the Antwerp University Hospital (UZA) has developed its own ERAS protocol for minimal-invasive lung surgery. The standard technique for this protocol is single-shot intercostal nerve blockade (ICNB) with ropivacaine.

This study wants to evaluate single-shot ICNB with ropivacaine versus ICNB with cryotherapy. Single-shot peripheral nerve blockade has a risk for increased need for opioids and less patient satisfaction compared to a continuous infusion technique, especially when using a multi-port robotic technique [6]. On the other hand, the technique is good in the majority of cases, easy to perform, low costs compared to the standard TEA care [7] and there is a lower incidence of adverse events [8]. Unilateral regional techniques are not associated with patient immobilisation, bladder dysfunction and hypotension [9]. The ICNB with cryotherapy is a newer technique with the advantage of blocking post-surgical pain for 1 to 3 months, while allowing the axons to regenerate. The risk for additional medication is therefore less. However, the disadvantage is the fact that the probes developed to induce this block are expensive and not refunded in Belgium. For this small randomized pilot study, 3 cryotherapy probes are given for free by the company AtriCure. This offers us the opportunity to study the outcome of ICNB with cryotherapy and ropivacaine (standard technique).

Postoperative pain that is not effectively treated or controlled will lead to chronic pain which is hard to control. Because of this it is really important to have an effective strategy in the first 3 months post-op to reduce chronic pain [10, 11]. With this study the investigators want to compare 2 techniques to see which analgesic single-shot technique meets the patient's satisfaction and it will also determine the most cost-effective pain strategy. When ICNB with cryotherapy seems promising compared to ICNB with ropivacaine in terms of patient satisfaction and pain control, a larger trial can be initiated.

The results of this study will give the investigators a first idea whether ICNB with cryotherapy can offer a clear advantage over ICNB with ropivacaine.

References

1. J. Hermanides, M.W. Hollmann, M.F. Stevens, P. Lirk. Failed epidural: causes and management. British Journal of Anaesthesia 109 (2): 144-54 (2012) 2. N. T. Ventham, M. Hughes, S. O'Neill, N. Johns, R. R. Brady and S. J. Wigmore. Systematic review and meta-analysis of continuous local anaesthetic wound infiltration versus epidural analgesia for postoperative pain following abdominal surgery. British Journal of Surgery 2013; 100: 1280-1289 4. A. Clemente, F. Carli. The physiological effects of thoracic epidural anesthesia and analgesia on the cardiovascular, respiratory and gastrointestinal systems. Minerva Anestesiologica 2008; 74: 549-63.

5. Timothy J.P. Batchelor, Neil J. Rasburn, Etienne Abdelnour-Berchtold, Alessandro Brunelli, Robert J. Cerfolio, et al. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERASVR) Society and the European Society of Thoracic Surgeons (ESTS). European Journal of Cardio-Thoracic Surgery 55 (2019) 91-115.

6. Ann E Bingham , Rochelle Fu, Jean-Louis Horn, Matthew S Abrahams. Continuous peripheral nerve block compared with single-injection peripheral nerve block: a systematic review and meta-analysis of randomized controlled trials. Reg Anesth Pain Med, Nov-Dec 2012;37(6):583-94.

7. Melissa Medina, Shannon R. Foiles, Matilde Francois, Carl V. Asche, Jinma Ren. Comparison of cost and outcomes in patients receiving thoracic epidural versus liposomal bupivacaine for video-assisted thoracoscopic pulmonary resection. The American Journal of Surgery 217 (2019) 520e524.

8. Marzia Umari, Stefano Falini, Matteo Segat, Michele Zuliani, Marco Crisman. Anesthesia and fast-track in video-assisted thoracic surgery (VATS): from evidence to practice. J Thorac Dis 2018;10(Suppl 4):S542-S554.

9. Alieh Zamani Kiasari, Anahita Babaei, Abbas Alipour, Shima Motevalli, Afshin Gholipour Baradari. Comparison of Hemodynamic Changes in Unilateral Spinal Anesthesia Versus Epidural Anesthesia Below the T10 Sensory Level in Unilateral Surgeries: a Double-Blind Randomized Clinical Trial. Med Arch. 2017 AUG; 71(4): 274-279 10. Blichfeldt-Eckhar M.R., Andersen, C., Ørding, H., Licht, P.B. & Toft, P. (2018). From acute to chronic pain after thoracic surgery: the significance of different components of the acute pain response. J Pain Res 11:1541-8. doi: 10.2147/JPR.S161303. PMID: 30147358; PMCID: PMC6101742.

11. Gan, T.J. (2017). Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res, 10:2287-98. doi:10.2147/JPR.S144066. PMID: 29026331; PMCID: PMC5626380.

ELIGIBILITY:
Inclusion Criteria:

Adult patients of 18 years or older who are able to give informed consent and fill out questionnaires in Dutch.

Exclusion Criteria:

* Patients who need an anatomic resection of the lung that's larger than one lung lobe, who have CPAM or infections.
* Patients with chronic use (>3 months) of strong opioids because of co-morbidities -for example, the use of tramadol is allowed.
* If there's a high risk of conversion to a thoracotomy. This will be evaluated by the lung surgeon.
* Patients who have had thoracic surgery in the past.
* Patients with chronic kidney disease stage 4 or 5 (GFR < 30 mL/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for anatomical lung resection (lobectomy or segmentectomy) with the intention of performing it by robotic-assisted thoracoscopic surgery (RATS) are eligible for the trial.
Sampling Method: Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The NRS pain score | Baseline, post-operative (day 0) in the recoveryward when the patient is awake and after 6 hours. Day 1-2-3 the NRS wil be measured in the morning, afternoon and evening. During the Follow-up visits: 2 weeks and 12 weeks after surgery
  The NRS score will be used to measure pain scores and this will be the primary outcome of the study.

SECONDARY OUTCOMES:
QoR-15 questionnaire | Measured at baseline, post-operative after surgery day 0, day 1, day 2 day 3 and day 4 during hospitalisation. At Folluw-up visit after 2 weeks and after 12 weeks
  The QoR-15 will provide a continuous variable with a minimum score of 0 and a maximum score of 150 and contains the most relevant questions concerning 5 domains (emotional status, physical comfort, psychological support, physical independence and pain) of overall well-being and recovery after surgery.
Lenght of stay | From date of hospitalization until discharge, estimated time of hospitalisation is 5 days, but we will measure until discharge from the hospital.
  Lenght of stay, defined as the total number of days in hospital after the surgical intervention.
Use of pain medication | during the postopertieve hospotalization periode, day 0 till day 3
  Cumulative use of systemic opioids and analgesics
Pain during mobilization | During the postopertieve hospotalization periode, day 0 till day 3
  Proportion of postoperative pain scores of NRS >3 during mobilization
Patient satisfaction | During post-opertieve periode day 0 - day 3.
  Measured using a likert 5-point scale going from Very unsatisfied to very satisfied.
Chest tube days | During post-opertieve periode day 0 - day 3, while hospilized.
  Time to removal of the chest tube in days;
urinary catheter in situ days | During post-opertieve periode day 0 - day 3, while hospilized.
  Time to removal of urinary catheter in days;
Degree of mobility | During post-opertieve periode day 0 - day 3, while hospilized.
  Degree of mobility (1-4 scale) at POD 1-3:
  1. on the bed
  2. to the chair
  3. to the toilet
  4. outside the patient's hospital room
  At POD 0 the degree of mobility is based on 2 options: patient hasn't been out of bed or went from bed to chair.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. J. Hendriks, MD. PhD., Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided